CLINICAL TRIAL: NCT02371161
Title: A Phase II Prospective Study of High-dose Myeloablative Therapy, With Stem Cell Devices Support in Elderly Patients (≥65 and ≤ 75 Years) With Relapsed Aggressive Non-Hodgkin Lymphoma or Resistant to First Line Therapy
Brief Title: Phase II of High-dose Therapy in Elderly Patients With Relapsed Aggressive NHL or Resistant to First Line Therapy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione Italiana Linfomi - ETS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FIL_RecAnz
Record Dates: First submitted 2015-02-11; First posted 2015-02-25 (Estimated); Last update posted 2018-04-25 (Actual); Status verified 2018-04

CONDITIONS: Non Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- R-DHAP/R-ICE (Experimental): High-dose myeloablative therapy (R-DHAP or R-ICE) and conditioning therapy (BEAM or FEAM) in elderly patients with relapsed NHL or resistant to firs line therapy
  Interventions: Drug: R-DHAP/R-ICE

INTERVENTIONS:
Drug: R-DHAP/R-ICE — R-DHAP/R-ICE 3 cycles every 21 days:
  1. R-DHAP
     * Rituximab 375 mg/m2, e.v. day 1
     * Desamethasone 40 mg days 1-4
     * cis-Platino100 mg/m2, day 2 (if ≥70 years 75 mg/m2)
     * Aracytin 2000 mg/m2, e.v. day 3 (if ≥70 years 1500 mg/m2)
  2. R-ICE
     * Rituximab 375 mg/m2, e.v. day 1
     * Etoposide 100 mg/mq, e.v. days 1,2,3 (if ≥70 years 75 mg/mq)
     * Ifosfamide with Mesna equidone 5000 mg/mq, day 2 (if ≥70 years 3750 mg/mq)
     * Carboplatino AUC=5, e.v. (max 800 mg/mq), day 2 (if ≥70 years AUC=4)
  Conditioning BEAM or FEAM
  Other Names: R-DHAP or R-ICE and BEAM or FEAM

SUMMARY:
A phase II prospective, non-randomized study. The study aim is to evaluate the feasibility and activity of high-dose therapy with stem cell in elderly patients with aggressive lymphoma relapsed FIT or resistant to first line therapy.

DETAILED DESCRIPTION:
The study aim is to evaluate the toxicity and activity of a therapeutic approach to high doses with support of peripheral blood stem cells (PBSC) in patients aged ≥ 65 and ≤75 years, chemosensitive relapsed or refractory to therapy first line in terms of event free survival (EFS) and treatment related mortality (TRM)

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of NHL
* relapse and refractory pts
* age ≥ 65 and ≤75
* ECOG performance status <2
* FIT patients (Instrumental Activity of Daily Living (IADL)=8, Activity of Daily Living (ADL)=6, Cumulative Illness Rating Scale (CIRS) =0 SCORE=3-4, <5 SCORE=2 )
* evaluable disease
* no RT since 3 week
* absolute neutrophil count >= 1500/mm3 and platelets >= 100.000/106L
* Creatinin <= 1.5 mg/dL and clearance >40 ml/min/24 h
* bilirubins < =2 mg/dL
* forced expiratory volume >50% - arterial pressure O2 >70 mmHg
* no other neoplastic disease
* Life expectancy> 3 months
* signed informed consent

Exclusion Criteria:

* HBV+ - HCV+ - HIV+
* NSC involvement - medullar infiltration > 20%
* other chemotherapy or radiotherapy
* cardiac disease
* alteration of liver and kidney function
* infections
* demented patient
* no compliance and depressed pts
* Frail and Unfit pts

Ages: 65 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 135 (Estimated)
Dates: Start 2014-02 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
Event free survival EFS | 36 months
  Evaluate the toxicity and activity of a therapeutic approach to high doses with stem cell support device (PBSC) in patients aged ≥ 65 and ≤75 years, chemosensitive relapsed or refractory to 1st line therapy in terms of EFS.
Treatment related mortality TRM | 100 days from the high doses
  Evaluate the toxicity and activity of a therapeutic approach to high doses with stem cell support device (PBSC) in patients aged ≥ 65 and ≤75 years, chemosensitive relapsed or refractory to 1st line therapy in terms of TRM.

SECONDARY OUTCOMES:
Complete Remission (CR) rate | 48 months (at the end of therapy)
Overall Survival (OS) | 48 months (at the end of therapy)
Adverse events incidence evaluation (grade III or IV) | 48 months (at the end of therapy)
  Number of participants with adverse events (grade III or IV)
Quality of Life (QoL) | 54 months
  Evaluate the quality of life (QoL) before, after therapy rescue and after six months of high-dose therapy through the quality of life questionnaire of European Organization for Research and Treatment of Cancer (EORTC QLQ-C30)
Immunologic evaluation | 54 months
  Rating basic immunology and 6 months after therapy high doses (lymphocyte subpopulations and Ig subclasses)

CONTACTS AND LOCATIONS:
Overall Officials: Luca Castagna, MD, Principal Investigator — IRCCS Humanitas
Locations (27):
- Italy (27):
  - A.O. SS.Antonio e Biagio e C. Arrigo, Alessandria, AL
  - Ospedali Riuniti, Ancona, AN
  - Ospedale Perrino, Brindisi, BR
  - Spedali Civili, Brescia, BS
  - Policlinico Vittorio Emanuele, Catania, CT
  - Casa Sollievo della Sofferenza, San Giovanni Rotondo, FG
  - IRST Meldola, Meldola, Forlì-Cesena
  - IRCCS San Martino - IST, Genova, GE
  - ASUR Marche, Area Vasta 3, Civitanova Marche, MC
  - AO Riuniti Papardo Piemonte, Messina, ME
  - IRCCS Humanitas, Rozzano, Milano
  - AO Niguarda Ca' Granda, Milan, MI
  - Ospedale Civile "Guglielmo da Saliceto", Piacenza, PC
  - Centro di Riferimento Oncologico, Aviano, PN
  - Azienda Ospaliero Universitaria di Parma, Parma, PR
  - Ospedale San Carlo, Potenza, PZ
  - AUSL di Ravenna, Ravenna, RA
  - A.O. Bianchi - Melacrino - Morelli, Reggio Calabria, RC
  - Asmn-Irccs, Reggio Emilia, RE
  - Policlinico Sant'Andrea, Roma, RM
  - Ospedale Nocera- Pagani, Nocera Inferiore, SA
  - AOU San Giovanni e Ruggi, Salerno, SA
  - AOU Città della Salute e della Scienza, Torino, TO
  - Ospedale Mauriziano, Torino, TO
  - AO Santa Maria, Terni, TR
  - Ospedale S.Andrea, Vercelli, VC
  - Ospedale degli Infermi, Rimini

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Tucci A, Re A, Pagani C, Marcheselli L, Marcheselli R, Malaspina F, Cavallo F, Zilioli VR, Zanni M, Mannina D, Michieli M, Arcari A, Castagna L, Musuraca G, Clerico M, Merli F, Tani M, Re F, Gini G, Rotondo F, Turrini M, Rossi G, Cox MC. A phase 2 study of autologous stem cell transplantation as salvage therapy for older patients with aggressive B-cell lymphoma prospectively evaluated by comprehensive geriatric assessment: the FIL_RECANZ study. Leuk Lymphoma. 2025 Jul;66(7):1284-1292. doi: 10.1080/10428194.2025.2471499. Epub 2025 Mar 8. PMID 40055982